CLINICAL TRIAL: NCT06205472
Title: Phase II Study of Adjuvant Simultaneously Integrated Boost Radiotherapy Following Narrow-Margin Hepatectomy in Patients With HCC.
Brief Title: Phase II Study of Adjuvant SIB Radiotherapy Following Narrow-Margin Hepatectomy in Patients With HCC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4255
Record Dates: First submitted 2023-12-25; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma; Narrow Margin; Radiotherapy
Keywords: Hepatocellular Carcinoma; Narrow Margin; Adjuvant Simultaneously Integrated Boost Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant SIB radiotherapy (Experimental): Adjuvant integrated boost radiotherapy following narrow-margin hepatectomy in patients with HCC.
  Interventions: Radiation: Adjuvant SIB radiotherapy

INTERVENTIONS:
Radiation: Adjuvant SIB radiotherapy — Eligibility patients will receive IMRT or VMAT to high risk area of tumor bed and tumor bed. The prescription dose to 95% GTVtb boost was planned at 55-60Gy, with PTV 45-50Gy, in 23-25 fractions,mainly depending on the dose constraints of OARs.

SUMMARY:
This is a single-arm prospective phase II clinical trial to investigate the efficacy and safety of adjuvant simultaneouslyintegrated boost radiotherapy following narrow-margin(<1cm) hepatectomy in patients with HCC. Eligibility patients will receive IMRT or VMAT to high risk area of tumor bed and tumor bed. The prescription dose to 95% GTVtb boost was planned at 55-60Gy, with PTV 45-50Gy, in 23-25 fractions, mainly depending on the dose constraints of OARs. The primary endpoint is the 3-year OS, the secondary endpoints are disease-free survival, patterns of failure, toxic events and local control rate.

DETAILED DESCRIPTION:
Surgical resection is the primary treatment for HCC. However, it is associated with a high rate of recurrence and death. Based on the results of our retrospective study and phase II study, adjuvant radiotherapy is an effective, tolerable, and promising adjuvant regimen in patients with narrow-margin(<1cm) after hepatectomy. The 3-year and 5-year OS rates of 88.2% and 72.2% were significantly higher than the expected rates based on published reports and exceeded our predetermined threshold. However, there is no standard for the prescription dose. The high risk area of recurrence is mostly close to the blood vessels in the tumor bed, and simultaneously integrated boost (SIB) technique can optimize the target dose while protecting normal tissues. So, the investigators conducted this single-arm prospective phase II clinical trial to investigate the efficacy and safety of adjuvant SIB radiotherapy following narrow-margin(<1cm) hepatectomy in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of HCC after hepatectomy with narrow pathological margins (< 1 cm)
* Age > 18 years
* Recovery from surgery with an Eastern Cooperative Oncology Group performance status score of 0 or 1
* Child-Push Score: A5-A6
* Estimated life expectancy > 3 months
* No distant metastasis (M0)
* Blood routine examination: Hb≥80g/L, ANC≥1.0x10^9/L, PLT≥50x10^9/L
* Hepatic function: alanine transaminase(ALT) and aspartate transaminase(AST) ≤1.5 times ULN; or ALT ≤ULN and AST ≤6 times ULN exclude possibility of heart disease
* Renal function: creatinine(CRE) and blood urea nitrogen(BUN)≤1.5 times ULN
* Voluntary to participate and sign informed consent

Exclusion Criteria:

* History of malignancies, except for basal cell skin carcinoma and in situ carcinoma of the cervix
* Had prior abdominal irradiation
* Had prior liver transplantation
* Had serious myocardial disease or renal failure
* Had moderate or severe ascites with obvious symptoms
* Duration from surgery ≥ 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-26 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
The 3-year Overall Survival | up to 36 months
  The 3-year overall survival was calculated from the date of surgical resection to the date of death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | up to 36 months
  Disease-free survival (DFS) was calculated from the date of surgical resection to the date of the first recurrence or death from HCC
Pattern of Failure | up to 36 months
  The type of recurrence (locoregional failures or distant failure)
Toxic Events | up to 36 months
  Toxic events was evaluated during received protocol therapy according to CTCAE 4.03
Local Control Rate | up to 36 months
  Patients with stable disease [SD], partial response [PR] or complete response[CR] were recorded as local control.

CONTACTS AND LOCATIONS:
Locations (1):
- Bo Chen, Beijing, China